CLINICAL TRIAL: NCT04273490
Title: Characterising Pain, Quality of Life, Body Composition, Arterial Stiffness, Muscle Function, Bone Density and Geometry in Adult Persons With Hereditary Hypophosphatemia and Healthy Controls
Brief Title: Characterising Pain, QoL, Body Composition, Arterial Stiffness, Muscles and Bones in Adult Persons With XLH and Healthy Controls
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 1107214219
Record Dates: First submitted 2019-11-05; First posted 2020-02-18 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-05

CONDITIONS: X-linked Hypophosphatemia; Hereditary Hypophosphatemia
MeSH Terms: conditions — Familial Hypophosphatemic Rickets

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum, white cells, urine, and bone tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hereditary hypophosphatemia: Adult persons with genetically or biochemically verified hereditary hypophosphatemia.
- Control: Adult control persons without disturbances in calcium, vitamin D or phosphate homeostasis matched on age, gender and menopausal status.

SUMMARY:
Hereditary hypophosphatemia (XLH) is a rare, inherited disease. Loss-of-function mutation in the phosphate regulating gene with homologies to endopeptidases on the X-chromosome (PHEX) results in excess fibroblast growth factor 23 (FGF23) production and manifests as rickets in children and osteomalacia in adults.

This study aims to characterize and measure pain, quality of life, muscle function, body composition, arterial stiffness, bone mineral density, geometry and microarchitecture in patients with XLH compared to age and gender-matched controls.

DETAILED DESCRIPTION:
Hereditary hypophosphatemia (XLH) is a rare, inherited disease. Loss-of-function mutation in PHEX results in excess fibroblast growth factor 23 (FGF23) production and manifests as rickets in children and osteomalacia in adults. FGF23 is a hormone that reduces renal phosphate reabsorption, decreases renal 1α-hydroxylase activity and increases renal 24-hydroxylase activity. As a consequence, individuals with XLH display hypophosphatemia and inadequate levels of 1,25(OH)2D (1). Therefore, conventional medical treatment of XLH aims to replace the loss with oral phosphate and activated vitamin D analogues.

The pain experienced by patients with hypophosphatemic rickets is not well characterized and needs to be addressed in order to establish the most optimal pain management in patients with XLH. The causes of pain experienced by patients with XLH are numerous: osteomalacia, enthesopathy, muscular pain, lower limb deformities, secondary arthrosis, nerve compression, and dental abscesses (3).

Quality of life (QoL) in patients with XLH is only briefly studied (4, 5). A French study found significantly decreased QoL among adult patients with XLH compared to patients with axial spondylarthritis. Especially enthesopathies were associated with a decreased QoL (4).

Increased blood levels of FGF23 are not associated with increased risk of cardiovascular disease in itself (6-8). However, conventional therapy for patients with XLH may increase their cardiovascular risk since complications to the therapy such as nephrocalcinosis and hyperparathyroidism are associated with increased cardiovascular risk. Arterial stiffness may be a valuable marker of increased cardiovascular risk as it has been able to predict cardiovascular disease and mortality in different populations (10, 11). If conventional therapy increases the risk of cardiovascular morbidity and mortality, arterial stiffness may be increased among patients with XLH which may depend on treatment status (i.e., currently treated, currently non-treated, accumulated (years of) treatment and treatment naïve).

Patients with XLH often complain about muscle fatigue and exhaustion. Muscle function in XLH is thought to be compromised by chronic hypophosphatemia, but the effect of XLH on muscle function has only been briefly evaluated (12, 13).

There are no available reports on body composition in XLH adults, but body mass index (BMI) in XLH is increased compared to controls (14).

In previous studies, examinations by high resolution peripheral quantitative computed tomography (HRpQCT) have shown significantly larger total bone area in patients with XLH compared to individuals without XLH. However, patients with XLH have a reduced number of trabeculae and cortical thickness (15). These differences are seen regardless of treatment. When receiving conventional treatment, the cortical porosity is significantly elevated compared to patients with XLH who receive no treatment (17).

HYPOTHESES:

Primary null hypotheses:

* There is no difference in pressure pain threshold between groups.
* There is no difference in QoL between groups.
* There is no difference in arterial stiffness assessed by tonometry between groups.
* There is no difference in 24h blood pressure between groups.
* There is no difference in muscle strength and function between groups.
* There is no difference in body composition between groups.
* There is no difference in bone mineral density, geometry, microarchitecture or estimated strength between groups.
* There is no difference in presence of osteoid-volume, -surface or -thickness, osteoclast number, osteoblastic surface, osteoblast morphology or mineralization time between groups.
* Osteomalacia is not more common in bone biopsies from patients with XLH compared to controls.

Secondary null hypotheses:

* There is no difference in arterial stiffness within the XLH group when stratifying for treatment status.
* There is no difference in 24h blood pressure within the XLH group when stratifying for treatment status.
* There is no difference in bone mineral density, geometry, microarchitecture or estimated strength within the XLH group when stratifying for treatment status.

MATERIALS AND METHODS

Study design:

A cross-sectional study of adult persons with XLH and an age- and gender-matched control group.

Population:

The investigators plan to include 50 persons with XLH and 50 control persons without disturbances in the calcium, vitamin D or phosphate homeostasis, matched by age (+/- 2 years) and gender. For women, matching will also be performed on menopausal status.

EXAMINATIONS

Questionnaires:

Pain will be assessed by a bone-specific questionnaire (FACT-BP), a questionnaire for general pain (Brief Pain Inventory (BPI)), and one for assessment of neuropathic pain (painDETECT).

The participant's level of catastrophic thinking will be assessed with the Pain Catastrophizing Scale (PCS). Depression and anxiety will be assessed with the Patient Health Questionnaire (PHQ-9) and Generalized Anxiety Disorder 7 (GAD-7).

Quality of Life will be measured by the SF-36 questionnaire (SF36v2).

Pressure algometry:

Mechanical pressure pain over the bone will be determined as force (N) per skin area (cm2) by a handhold pressure algometer with a 1 cm2 probe (Algometer II, Somedic SenseLab AB) (18). The 1 cm2 probe will be directed perpendicularly to the skin and pressure will be applied at a constant force increase rate until the participant identifies the pressure as pain and presses a button (pressure pain threshold (PPT)). PPT will be measured over the sternum and also corresponding to the tibia 5 cm below the patella. The skin between the thumb and the index finger of the non-dominant hand will be measured as a control site.

Biochemistry:

Blood samples will be collected in a fasting state. The investigators will measure ionized calcium, phosphate, magnesium, creatinine, parathyroid hormone (PTH), vitamin D metabolites (such as 25OHD; 1,25(OH)2D; 24,25(OH)2D; 1,24,25(OH)3D), vitamin D binding protein, FGF23, sclerostin, Klotho, osteopontin, and bone turnover markers (such as CTX, P1NP, osteocalcin and bone-specific alkaline phosphatase), and relevant genes for hereditary hypophosphatemia (if not previously genetically verified).

24 hour urine will be collected for measurement of calcium, phosphate, magnesium, creatinin, sodium and potassium.

Blood pressure and arterial stiffness 24-hour blood pressure will be measured using Arteriograph24. Arterial stiffness and pulse wave analysis (PWA) will be assessed by tonometry using the SphygmoCor system (Xcel; AtCor Medical, Sydney, NSW, Australia). Participants treated with betablockers will be excluded from blood pressure and arterial stiffness measurements.

Muscle function The investigators will assess upper and lower extremity strength by handgrip strength, elbow flexion and extension, and knee flexion and extension using the adjustable dynamometer chair (Good Strength; Metitur Ltd, Finland). To assess physical function, the investigators will use the Timed Up and Go (TUG) test, repeated chair rising, repeated weight lifting and 6-minutes' walk test (6 MWT).

Physical examination In order to quantify the degree of malformation of the joints in the lower extremities, the smallest distance between knees and between ankles will be measured in standing, weight bearing position.

Joint mobility The investigators will assess joint function in enthesopathy-suspected joints (neck/back, hip, knee and ankle) as well as shoulder, elbow, wrist and knee in order to discriminate between pain originating from osteomalacia or from enthesopathies.

Body composition and VFA using DXA Body composition and bone mineral density (Forearm, hip, lumbar spine and whole body) will be assessed by dual energy X-ray absorptiometry (DXA) (Discovery A scanner; Hologic, USA). Obtaining vertebral fracture assessment (VFA) by DXA enables us to exclude reported back pain being due to vertebral compression fractures.

High-resolution peripheral Quantitative Computed Tomography:

A HRpQCT bone scan of the dominant distal tibia and radius will be performed using an Xtreme CT-scanner (SCANCO Medical AG, Switzerland).

Bone biopsies:

Optional bone biopsies will be taken after assessment of pain characteristics. Participation in the overall study is allowed without participating in this examination.

One 7 mm biopsy marked with tetracyclin 14, 13, 4, and 3 days prior will be fixed in ethanol and analysed by HRpQCT, Nano-scale and histomorphometry.

ELIGIBILITY:
Inclusion Criteria:

* Understand oral and written Danish
* Able to consent

For XLH only:

1. genetically verified XLH by detection of a disease-causing mutation in PHEX or a positive family history of X-linked hypophosphatemia.
2. biochemically verified hereditary hypophosphatemia: serum PO4 below normal range and low TmPO4/GFR, and/or elevated serum FGF23 and a history of childhood rickets or spontaneous endodontic abscesses to exclude acquired hypophosphatemia, e.g., tumor-induced osteomalacia.

   Exclusion Criteria:
   * P-25OHD < 25 mmol/L*
   * Severe co-morbidities, which in the opinion of the investigator may have major impact on study outcomes. This may include, but is not limited to o poorly controlled hyperthyroidism o Paget disease

     o type 1 diabetes mellitus or poorly controlled type 2 diabetes mellitus

     o severe and chronic cardiac, liver, or renal disease

     o Cushing syndrome

     o Rheumatoid arthritis

     o Active pancreatitis

     o Malnutrition

     o Recent prolonged immobility*

     o Active malignancy (including myeloma)
   * Treatment with

     o Burosumab
     * Beta-blockers
     * Oral steroids
   * For controls only:

     * disturbances in the calcium or phosphate homeostasis

       * participants with low 25OHD levels or recent immobility may be re-screened for participations 6 months after this has been corrected

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 persons with hereditary hypophosphatemia and 50 control persons without disturbances in the calcium, vitamin D or phosphate homeostasis, matched by age (+/- 2 years) and gender. For women, matching will also be performed on menopausal status (pre-, peri-, and postmenopausal*).
  *Pre-menopausal = regular periods Peri-menopausal = irregular periods +/- hot flashes Post-menopausal = last period ≥1 year ago
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
PPT | Day 2
  Pressure pain threshold assessed by pressure algometry
Quality of life in patients with bone-specific pain | Day 1
  Assessed by questionnaire (FACT-BP) on a scale from 0 to 4. Higher scores mean a worse outcome.
General pain: Brief Pain Inventory | Day 1
  Assessed by questionnaire (Brief Pain Inventory) on a scale from 0 to 10. 0 meaning no pain, 10 meaning worst pain ever.
Neuropathic pain: questionnaire (painDETECT) | Day 1
  Assessed by questionnaire (painDETECT) on a scale from 0 to 10. 0 meaning no pain, 10 meaning worst pain ever.
Health-related quality of life: SF36v2 | Day 1
  Assessed by questionnaire (SF36v2) on a scale from 1 to 5. Higher scores meaning a worse outcome.
Systolic and diastolic blood pressure | 24 hours
  24 hour blood pressure of the upper right arm
Pulse wave velocity | 45 minutes
  Assessed by tonometry using SphygmoCor system
Arterial stiffness | 45 minutes
  Assessed by tonometry using SphygmoCor system
Arterial stiffness | 24 hours
  Assessed by tonometry using Arteriograph24
Maximum strength | Day 2
  Handgrip strength, elbow and knee flexion and extension assessed by dynamometer chair (Good Strength; Metitur Ltd, Finland).
Maximal force production | Day 2
  Handgrip strength, elbow and knee flexion and extension assessed by dynamometer chair (Good Strength; Metitur Ltd, Finland).
Timed Up and Go | Day 2
  Measures the time to stand up, walk three metres in a straight line, and immediately return to the chair.
Repeated chair rising | Day 2
  Measures the time for ten consecutive chair rises.
Repeated weight lifting | Day 2
  Measures the time for ten consecutive weight lifts.
6-minutes' walk test | Day 1
  Measures the distance walked in 6 minutes.
Body composition | Day 2
  Assessed by DXA
Vertebral Fracture Assessment | Day 2
  Assessed by DXA
Volumetric bone mineral density | Day 1
  Assessed by HRpQCT of distal tibia, distal radius, and bone biopsy
Bone geometry | Day 1
  Assessed by HRpQCT of distal tibia, distal radius, and bone biopsy
Bone microarchitecture | Day 1
  Assessed by HRpQCT of distal tibia, distal radius, and bone biopsy
Estimated bone strength | Day 1
  Assessed by HRpQCT of distal tibia, distal radius, and bone biopsy
Mineralization rate | 14 days
  Histomorphometry on bone biopsy
Mineralization lag time | 14 days
  Histomorphometry on bone biopsy
Osteoid volume | 14 days
  Osteoid volume in trabecular and compact bone assessed by histomorphometry on bone biopsy
Osteoid thickness | 14 days
  Osteoid thickness in trabecular and compact bone assessed by histomorphometry on bone biopsy
Osteoid surface covering | 14 days
  Osteoid surface covering in trabecular and compact bone assessed by histomorphometry on bone biopsy
Percentage of surface covered by osteoblasts | 14 days
  Assessed by histomorphometry on bone biopsy
Percentage of surface covered by osteoclasts | 14 days
  Assessed by histomorphometry on bone biopsy
Lacunar concentration of mineralization inhibitors | 14 days
  Assessed by nano-scale on bone biopsy

SECONDARY OUTCOMES:
Catastrophic thinking | Day 1
  Assessed by questionnaire (Pain Catastrophizing Scale) on a scale from 0 to 4. Higher scores mean a worse outcome.
Depression | Day 1
  Assessed by questionnaire (Patient Health Questionnaire) on a scale from 0 to 3. Higher scores mean a worse outcome.
Anxiety | Day 1
  Assessed by questionnaire (Generalized Anxiety Disorder 7) on a scale from 0 to 3. Higher scores mean a worse outcome.

OTHER OUTCOMES:
Smallest distance between knees. | Day 1
  Measured in standing, weight bearing position.
Smallest distance between ankles. | Day 1
  Measured in standing, weight bearing position.
Joint mobility | Day 1
  Passive mobility of the neck, shoulder, elbow, wrist, ankle, back, hip and knee will be measured from anatomic neutral position using a protractor and compared to normal values.
Areal bone mineral density (aBMD) | Day 2
  BMD at the lumbar spine, femoral neck and distal forearm assessed by DXA
Plasma concentration of ion-calcium | Day 1
  Plasma concentration of ion-calcium taken in a fasting state
Plasma concentration of phosphate | Day 1
  Plasma concentration of phosphate taken in a fasting state
Plasma concentration of magnesium | Day 1
  Plasma concentration of magnesium taken in a fasting state
Plasma concentration of creatinine | Day 1
  Plasma concentration of creatinine taken in a fasting state
Plasma concentration of PTH | Day 1
  Plasma concentration of PTH taken in a fasting state
Concentration of vitamin D metabolites | Day 1
  Plasma levels of 25OHD, 1,25(OH)2D, 24,25(OH)2D, 1,24,25(OH)3D and vitamin D-binding protein taken in a fasting state
Plasma concentration of FGF23 | Day 1
  Plasma concentration of FGF23 taken in a fasting state
Plasma concentration of sclerostin | Day 1
  Plasma concentration of sclerostin taken in a fasting state
Plasma concentration of klotho | Day 1
  Plasma concentration of klotho taken in a fasting state
Plasma concentration of osteopontin | Day 1
  Plasma concentration of osteopontin taken in a fasting state
Plasma concentrations of bone turnover markers | Day 1
  Plasma levels of bone-specific alkaline phosphatase, osteocalcin, procollagen type I N-terminal propeptide (P1NP), C-terminal telopeptide (CTX)
Plasma concentration of tissue non-specific alkaline phosphatase | Day 1
  Plasma levels of tissue non-specific alkaline phosphatase taken in a fasting state
Urine calcium | 24 hours
  24 hours urine calcium
Urine phosphate | 24 hours
  24 hours urine phosphate
Urine magnesium | 24 hours
  24 hours urine magnesium
Urine creatinine | 24 hours
  24 hours urine creatinine
Urine sodium | 24 hours
  24 hours urine sodium
Urine potassium | 24 hours
  24 hours urine potassium

CONTACTS AND LOCATIONS:
Overall Officials: Lars Rejnmark, Principal Investigator — Dept. of Endocrinology and Internal Medicine, The Osteoporosis Clinic
Locations (1):
- Dept. of Endocrinology and Internal Medicine, The Osteoporosis Clinic, Aarhus N, Denmark